CLINICAL TRIAL: NCT03803033
Title: Cost-benefit Analysis of a Clinical Pharmacist Intervention in Preventing Adverse Drug Events in the General Chronic Diseases Outpatients
Brief Title: Cost-benefit Analysis of a Clinical Pharmacist Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1IRB/2014/50
Record Dates: First submitted 2018-12-24; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Chronic Disease
Keywords: Treatment-related problems; Cost saving; Clinical pharmacy
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Chronic diseases patients were initially assigned to either 3 months of routine care service (control group) or to an experimental clinical pharmacy-based HMMR service (intervention group) in the outpatient clinic setting of the Jordan University Hospital in Amman, Jordan.
Who Masked: Participant
Masking Description: A prospective single-blind randomized control trial (RCT) for evaluating the economic impact of a clinical pharmacist's identifying and managing of TRPs as part of an home medication management review
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The objective of the group was to introduce an experimental clinical pharmacy-based home medication review service in the outpatient clinic setting of the Jordan University Hospital in Amman, Jordan. The intervention under evaluation in the study is the pharmacy-based home medication review service.
  Interventions: Other: Clinical pharmacy-based home medication management review service
- Control (No Intervention): The objective of the control group was to identify changes in treatment and associated costs that take place in patients as part of the usual practice, as compared to the intervention arm, regardless of the clinical pharmacist service intervention.

INTERVENTIONS:
Other: Clinical pharmacy-based home medication management review service — A baseline interview by the clinical pharmacist was conducted with patients at their homes to assess their use of treatment and to collect all relevant information needed to identify TRPs. Upon TRP identification at baseline, the clinical pharmacist generated a written report of findings and recommendations, which was delivered directly to the patient's physician in a sealed envelope. Patients were asked to refer back to their physicians if they required confirmation of any changes in treatment. Physicians maintained the blinding of patients with regard to whether changes were based on recommendations by the pharmacist. In both the intervention and the control groups, the clinical pharmacist performed a follow-up interview with patients 3 months after the initial interview, during a regular follow-up visit to their physician at the hospital. Assessments in the follow-up interview, regardless of the study group, involved changes in treatment and number of TRPs.
  Arms: Intervention

SUMMARY:
Clinical pharmacy services are vital in the prevention of adverse drug events (ADEs) in clinical practice, extending beyond the hospital to chronic disease management in outpatient settings. This study sought to evaluate the cost-benefit of a clinical pharmacy intervention in resolving treatment-related problems (TRPs) among hospital outpatients with chronic diseases. From the hospital system perspective, the cost-benefit analysis was based on a randomized clinical trial in the general outpatients of the major hospital in Jordan. Eligible patients were randomly assigned to either an intervention or a control group. TRPs were identified in both study groups, but interventions were delivered only to the intervention group via a home medication management review (HMMR) by a clinical pharmacist. A follow-up in both groups took place 3 months after recruitment. The total economic benefit was the sum of (i) cost savings due to intervention and (ii) cost avoidance associated with preventable ADEs. The primary outcome measures were the net benefit and benefit-to-cost ratio with the clinical pharmacist-based HMMR. Based on both of the annual net benefit and benefit-to-cost ratio, the study intervention demonstrated to be cost beneficial. Sensitivity analyses confirmed the robustness of results. The RCT-based cost-benefit evaluation provided evidence-based insight into the economic benefit of a clinical pharmacist-provided HMMR for preventing ADEs in the general chronic diseases outpatients. This intervention method against the TRPs among outpatients is cost beneficial and offers substantial cost savings to the healthcare hospital payer in Jordan.

DETAILED DESCRIPTION:
Economic evaluation The total economic benefit of the intervention was calculated as the sum of the cost savings and the cost avoidance associated with the intervention.

Cost savings Cost savings based on the intervention were the reduced cost of therapy associated with treatment changes due to the intervention. Cost savings were therefore calculated as (the reduced cost of therapy in the intervention arm) minus (the reduced cost of therapy in the control arm).

Cost avoidance Cost avoidance was the cost avoided by eliminating the occurrence of ADEs as a consequence of the pharmacist interventions.

* Based on the method of Nesbit et al., utilizing an expert panel of four specialist clinical pharmacists, the likelihood of an ADE in the absence of the intervention was set. The intervention with the potential to prevent an ADE was assessed for cost avoidance.
* The cost of an ADE was calculated on the assumption that an ADE in an outpatient will lead to a single admission to an internal medicine ward via an emergency department visit.
* For each intervention with the potential to prevent an ADE, cost avoidance was calculated by multiplying the probability of an ADE in the absence of the intervention (calculated via the Nesbit method) by the average cost of an ADE. The overall cost avoidance was the sum of avoided cost with all interventions for TRPs.

Cost-benefit analysis The net benefit was calculated as (cost saving) + (cost avoidance). It was assumed that no intervention would increase the probability of a preventable ADE.

* Calculating monthly cost savings and avoidance was based on a capacity on the part of the pharmacist to perform three HMMRs in a day, for an underestimated average of 21 working days a month, summing to a total of 63 patients per month. The need for a monthly outcome cost stems from the fact that outpatient pharmacists are paid monthly in Jordan. The assumption of three HMMRs per day is based on the expectation that a single home visit will last a maximum of 1 hour, as discussed earlier, and that up to 2 to 3 hours are needed to identify TRPs, write the physician letter, contact the physician, and implement the recommendations.
* The cost of the intervention was calculated as (the salary of a regular outpatient pharmacist) + (any increased cost of therapy in the intervention arm, measured as -ve cost saving). Here, the increased cost of therapy with intervention is referred to as '-ve cost saving' in contrast to +ve cost saving, which indicates the reduction in the cost of therapy because of treatment changes in the intervention group, as discussed above.
* The benefit-to-cost ratio was the (sum of cost savings and cost avoidance) divided by (cost of the intervention). The net benefit of the intervention was the (sum of cost savings and cost avoidance) minus (cost of the intervention).

Only direct medical costs were considered in calculations, and all costs were adjusted based on the Jordanian consumer price index to the financial year 2017/18.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* with at least one chronic disease, defined as a condition requiring prolonged management for a minimum of 3 months;
* living in Jordan for the past year;
* intention to remain in Jordan for the 3-month study duration;
* met at least one of the following criteria:
* taking ≥5 medications, taking ≥12 doses a day, discharged from the hospital within the past 4 weeks, exposed to significant changes in medication regimens within the past 3 months, demonstrating symptoms of potential adverse drug reactions, or demonstrating a poor therapeutic response to medication therapy. A significant change to medication regimen was defined as discontinuing a medication, starting new medications, or stepping up because of actual or potential therapy failure or guideline recommendations. A poor therapeutic response was defined as persistence of symptoms despite treatment.

Exclusion Criteria:

* Patients who don't have a chronic disease
* Cognitive or sensory impairment that may prevent conducting the interview
* Pregnant patients
* Patients who are planning to travel within the next 3 months after the baseline visit to the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cost-benefit analysis | Three months
  The benefit-to-cost ratio was the (sum of cost savings and cost avoidance) divided by (cost of the intervention). The net benefit of the intervention was the (sum of cost savings and cost avoidance) minus (cost of the intervention).
  The scope of this is limited to cost consequences of TRPs and interventions addressing them, and does not include humanistic and clinical outcomes of interventions. Net benefit and benefit-to-cost ratio with the clinical pharmacist-based home-based service.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Iman Basheti, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided